CLINICAL TRIAL: NCT06831383
Title: The STOP-HPV Scale Up Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Medical Group Association (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-000022; 1R01CA276151-01 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Human Papilloma Virus Vaccine
Keywords: Human Papillomavirus Vaccination; Practice-based improvement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STOP-HPV Online (Experimental): Provider communication training
  Interventions: Behavioral: STOP-HPV-Online
- STOP-HPV LC (Experimental): Provider communication training plus Learning Collaborative sessions attended by practice leads and quarterly performance feedback to the practice.
  Interventions: Behavioral: STOP-HPV-LC
- Usual Care (No Intervention): Standard of care control

INTERVENTIONS:
Behavioral: STOP-HPV-Online — Approximately one third of practices within a participating health system will be randomized to receiving the STOP-HPV-Online intervention.
  Arms: STOP-HPV Online
Behavioral: STOP-HPV-LC — Approximately one third of practices within a participating health system will be randomized to receiving the STOP-HPV-LC intervention.
  Arms: STOP-HPV LC

SUMMARY:
Human papillomavirus (HPV) causes 35,900 US cancer cases per year, 4,000 deaths, and $4 billion in can In this study, the investigators will conduct a 3-arm clustered randomized controlled trial (RCT) in an estimated 72 practices from up to 8 health systems to evaluate the effectiveness and cost effectiveness of two potentially scalable implementation strategies (based on prior work) to increase the initiation of HPV vaccine against a usual care (control) arm. The intervention arms are 1) online provider communication training only ("STOP-HPV-Online" and 2) online provider communication training plus a Learning Collaborative, with performance feedback, attended by practice leads ("STOP-HPV-LC).

cer-related costs. It is recommended at ages 11-12 years routinely but can be given starting at ages 9-10 years. Despite having an effective vaccine, HPV vaccine initiation/completion rates in the U.S. were only at 76.8%/61.4% respectively in 2023 among 13-17 year olds; these rates are lower than the other recommended adolescent vaccines. Two key barriers are 1) suboptimal clinician communication to address parental concerns and 2) ineffective office systems causing missed vaccine opportunities.

DETAILED DESCRIPTION:
In prior work, the investigators have tested two implementation strategies/interventions that were effective, but which were deployed by the research team. The first is provider communication training ("STOP-HPV-Online"), delivered by the research team, in a cluster RCT in 48 pediatric practices from a research network (6.8% improvement in initiation). The other is a quality improvement, pre-post study, that included both provider communication training, as well as a Learning Collaborative (LC) for practice leads (8% increase in initiation).

A major challenge in implementation science and spreading practice-based strategies is to move from research teams deploying implementation strategies (intervention) to health systems deploying them. In this study, the investigators will compare the effectiveness and cost-effectiveness of the two implementation strategies (interventions) using a 3-arm clustered RCT: 1) STOP-HPV-Online vs 2) STOP-HPV-LC vs 3) usual care. The study team will randomize an estimated 72 practices (from up to 8 health systems) to the 1) STOP-HPV-Online arm, 2) the STOP-HPV-LC arm or 3) the control arm, assess fidelity to the intervention and conduct the evaluation. A collaborating organization, AMGA (the American Medical Group Association), will facilitate training of the health system personnel, as needed; however, the health systems will deploy each intervention. The primary outcome measure is the initiation rate among 9-<13 year olds with a well-child care visit during the 12 month intervention period (with inclusion starting at the time of a well child care visit during the intervention period). A secondary outcome measure will be the initiation rate among 13-17 year olds with a well child care visit during the intervention period (with inclusion starting at the time of a well child care visit during the intervention period. For both measures, inclusion criteria will be: 1) presenting to a participating practice, 2) age eligible at the visit and 3) no prior vaccine at the time of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient of participating practice
* Well child care visit during the 12-month intervention period
* No prior dose of HPV vaccine at the time of the well child care visit
* Age-eligible

Exclusion Criteria:

* Prior dose of HPV vaccine

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Initiation (first dose) of HPV vaccination among 9-<13 year olds at or following a well care visit with a participating provider during the intervention period. | 12 months from start of intervention
  The percent of children ages 9-<13 years of age who received their first dose of HPV vaccine at or following a well child care visit with a participating provider during the intervention-period (denominator is children ages 9-<13 with a well child visit during the study period at which they were due for their first dose).

SECONDARY OUTCOMES:
Initiation (first dose) of HPV vaccination among 13-17 year olds at or following a well care visit with a participating provider during the intervention period. | 12 months from start of intervention
  The percent of children ages 13-17 years of age who received their first dose of HPV vaccine at or following a well child care visit with a participating provider during the intervention-period (denominator is children ages 9-<13 with a well child visit during the study period at which they were due for their first dose).
Initiation (first dose) of HPV vaccination among 9-<13 year olds at or following a well care visit with any provider during the intervention period. | 12 months from start of intervention
  The percent of children ages 13-17 years of age who received their first dose of HPV vaccine at or following a well child care visit with any provider (participating or not) during the intervention-period (denominator is children ages 9-<13 with a well child visit during the study period at which they were due for their first dose).
Initiation (first dose) of HPV vaccination among 13-17 year olds at or following a well care visit with any provider during the intervention period. | 12 months from start of intervention
  The percent of children ages 13-17 years of age who received their first dose of HPV vaccine at or following a well child care visit with any provider (participating or not) during the intervention-period (denominator is children ages 9-<13 with a well child visit during the study period at which they were due for their first dose).
Total implementation cost | 12 months from start of intervention
  The difference in costs between arms will be used to calculate the incremental cost-effectiveness ratio (ICER)